CLINICAL TRIAL: NCT05610332
Title: Clinical Efficacy of Albumin Paclitaxel Plus Carrelizumab Versus FLOT in Neoadjuvant Treatment of Locally Advanced Gastric Cancer With Different Immunotypes--A Multi-center, Randomised, Open, Phase 3 Clinical Trial
Brief Title: Clinical Efficacy in Neoadjuvant Treatment of Locally Advanced Gastric Cancer With Different Immunotypes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of gastric surgery, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Arise-FJ-G007
Record Dates: First submitted 2022-10-06; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immune activated experimental group (Experimental): Albumin paclitaxel 260mg/m2, ivgtt, d1, d8 Carrelizumab: 200mg, ivgtt, d1, q3w
  Interventions: Drug: Camrelizumab; Drug: Albumin Taxol
- Immune activated control group (Active Comparator): Docetaxel 50mg/m2, ivgtt, d1, q14d; Oxaliplatin 85mg/m2, ivgtt, d1, q14d; Calcium folinate 200mg/m2, ivgtt, d1, q14d; 5-fluorouracil 2600mg/m2, 24h civ, d1, q14d
  Interventions: Drug: FLOT scheme
- Immune silence experimental group (Experimental): Carrelizumab: 200mg, ivgtt, d1, q3w Docetaxel 50mg/m2, ivgtt, d1, q14d; Oxaliplatin 85mg/m2, ivgtt, d1, q14d; Calcium folinate 200mg/m2, ivgtt, d1, q14d; 5-fluorouracil 2600mg/m2, 24h civ, d1, q14d
  Interventions: Drug: Camrelizumab; Drug: FLOT scheme
- Immunosilent control group (Active Comparator): Docetaxel 50mg/m2, ivgtt, d1, q14d; Oxaliplatin 85mg/m2, ivgtt, d1, q14d; Calcium folinate 200mg/m2, ivgtt, d1, q14d; 5-fluorouracil 2600mg/m2, 24h civ, d1, q14d
  Interventions: Drug: FLOT scheme

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab One course will last 21 days. Given once every 3 weeks at a dose of 200 mg.
  Arms: Immune activated experimental group; Immune silence experimental group
Drug: Albumin Taxol — Albumin paclitaxel was administered intravenously (without pretreatment) for 30 min on the first day of each cycle
  Arms: Immune activated experimental group
Drug: FLOT scheme — Docetaxel 50mg/m2, ivgtt, d1; Oxaliplatin 85 mg/m2, ivgtt, d1; Calcium folinate 200mg/m2, ivgtt, d1; 5-fluorouracil 2600mg/m2, 24h civ, d1,
  4 cycles before and after operation, q2w
  Arms: Immune activated control group; Immune silence experimental group; Immunosilent control group

SUMMARY:
To evaluate the clinical efficacy of albumin paclitaxel combined with carelizumab and FLOT in the neoadjuvant treatment of locally advanced gastric cancer with different immune types

DETAILED DESCRIPTION:
Background: At present, there is still a lack of prospective data to systematically compare the clinical efficacy of different neoadjuvant therapies in patients with different genotypes. To explore the clinical efficacy and safety of albumin paclitaxel combined with carrelizumab compared with FLOT neoadjuvant therapy in patients with locally advanced gastric cancer of different immune types.

Methods: This study is a multi center prospective study. 216 patients with gastric adenocarcinoma were included in the study to explore the proportion of PD-L1 positive cells in tumor tissue, evaluate the expression of PD-L1, serum HBV DNA level or other biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years, all sex； 2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by histology or cytology； 3. CT/MRI,PET-CT or laparoscopic exploration were used to confirm the diagnosis of gastric cancer staging as cT2-4a and/or N+ and M0 before operation.； 4. Measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.（CT scan of tumor lesion length≥10mm，CT scan short diameter of lymph node≥15mm，scan slice thickness 5mm）; 5. ECOG(Eastern Cooperative Oncology Group) PS(Performance Status):0-1 scores; 6. The expected survival time is more than 12 weeks; 7. The main organ function is normal, which should meet the following criteria:

1. blood routine examination standards should be met（no blood transfusion within 14 days）

   1. HB≥100g/L，
   2. WBC≥3×109/L
   3. ANC≥1.5×109/L，
   4. PLT≥100×109/L；
2. biochemical examination shall comply with the following criteria：

   1. BIL <1.5normal upper limit（ULN），
   2. ALT和AST<2.5ULN，GPT≤1.5×ULN；
   3. serum Cr≤1ULN，creatinine clearance rate>60ml/min（Cockcroft-Gault formula） 8. women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug.； 9. No other clinical studies were conducted before and during the treatment； participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Previous history of chemotherapy, radiotherapy, targeted drug therapy or immunotherapy
2. Patients with contraindications for surgical treatment and chemotherapy or whose physical condition and organ function do not allow for major abdominal surgery；
3. Patients with metastasis；
4. Having any active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Patients with vitiligo or cured childhood asthma/allergies who did not need any intervention in adulthood were excluded; Autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone; Type 1 diabetes with stable doses of insulin；
5. A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation；
6. Accompanied by serious heart, lung, liver, kidney disease; Have nerve, mental disease; Jaundice or obstruction of the digestive tract with severe infection；
7. Pregnant or lactating women；
8. The blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg)；
9. With Ⅰ magnitude of coronary heart disease, arrhythmia (including QTc protracted between male > 450 ms, women > 470 ms) and cardiac insufficiency；
10. Patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency;；
11. Subjects have failed to control good cardiovascular clinical symptoms or disease, including but not limited to: such as: (1) the NYHA class II heart failure or above (2) unstable angina pectoris (3) MI occurred within 1 year (4) have clinical significance of supraventricular or ventricular arrhythmias without clinical intervention on or after clinical intervention is still poorly controlled；
12. History of interstitial lung disease (except radiation pneumonia without hormone therapy), and history of non-infectious pneumonia；
13. Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g)；
14. A person who has previously been allergic to any component of the drug in this study； The researchers consider those who were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 4 months
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

SECONDARY OUTCOMES:
R0 resection rate | 4 months
  The surgical procedure was total or subtotal gastrectomy with 3 weeks after total neoadjuvant therapy
Disease control rate | 4 months
  Disease control rate
1-year and 3-year OS | 1 and 3 years
  1-year and 3-year OS
1-year and 3-year DFS | 1 and 3 years
  1-year and 3-year DFS
Adverse event | 3 years
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery
30 days mortality rates | 30 days
  Defined as the event observed within 30 days after surgery
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course
The prediction performance of Exosome contents (including proteins, nucleic acids) | 3 years
  Exosomes were isolated using a Backman Optima XPN-100 instrument. The exosomes morphology was characterized using a HT7700 transmission electron microscope (Hitachi, Co. Ltd., Japan). Fluorescent spectra were recorded using a F96 Pro fluorospectrophotometer (Shanghai Lengguang Technology). The concentration and size distribution of the exosomes were quantified using nanoparticle tracking analysis (NanoSight NS 300, Malvern Instrument). The obtained results were subjected to biostatistical analysis, such as heat map generation, ROC curve establishment, and confusion matrix.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Ph.D., Principal Investigator — Fujian Medical University Union Hospital
Locations (2):
- China (2):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Department of Gastric Surgery, Fuzhou, Fujian